CLINICAL TRIAL: NCT05229120
Title: Improving Delay Discounting to Decrease Harsh Parenting Among Parents Receiving Substance Use Treatment in Low Income Community
Brief Title: Improving Delay Discounting to Decrease Harsh Parenting Among Parents Receiving Substance Use Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: University of Maryland, College Park (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Julia Felton, Assistant Scientist, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NAP: 14781-29
Record Dates: First submitted 2022-01-18; First posted 2022-02-08 (Actual); Results first posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-02

CONDITIONS: Behavioral Health
Keywords: episodic future thinking; delay discounting; parent-child relations; low income; substance use treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Episodic Future Thinking (Experimental): Parents who are receiving residential substance use disorder (SUD) treatment will receive an adapted episodic future thinking focused condition. Parents will meet with peer recovery coaches (PRCs) who will administer the intervention, focused on generating future, pleasant events with their children. After the intervention session, parents will receive a daily postcard over the course of two weeks including a reminder cue generated as part of the episodic future thinking (EFT) intervention and a prompt to remember these episodes in vivid detail.
  Interventions: Behavioral: Episodic Future Thinking

INTERVENTIONS:
Behavioral: Episodic Future Thinking — The adapted episodic future thinking (EFT) intervention will focus on generation of vivid, substance-free, rewarding events that could happen in the future with their children.

SUMMARY:
Parents with substance use disorders are disproportionately more likely to engage in harsh physical discipline, which can lead to serious clinical outcomes, including child maltreatment and the intergenerational transmission of addictive disorders. One mechanism linking substance use and maladaptive parenting strategies is parental delay discounting, or the tendency to value smaller, immediate rewards (such as stopping children's misbehavior via physical punishment) relative to larger, but delayed rewards (like shaping adaptive child behaviors over time). This study will examine the efficacy of implementing a low-cost, brief intervention targeting the reduction of parental delay discounting to inform broader public health efforts aimed at reducing child maltreatment and interrupting intergenerational cycles of substance abuse in traditionally underserved communities.

DETAILED DESCRIPTION:
Parents with substance use disorders (SUD) are significantly more likely to engage in harsh parenting practices, including spanking, hitting, and belittling their children, than parents without SUD. Punitive physical and emotional discipline is, in turn, associated with increased rates of child maltreatment and the subsequent intergenerational transmission of substance use disorders. Parents in residential substance use treatment facilities are among those at highest risk for perpetrating harsh and abusive parenting; yet most behaviorally based parenting interventions available within inpatient settings do not take into account the unique mechanisms linking parental substance use to harsh parenting. Specifically, parents with SUD may be at heightened risk for engaging in maladaptive parenting approaches given a tendency to prioritize immediate rewards (such as stopping a child's misbehavior using physical punishment) relative to larger, but delayed rewards (including shaping positive child behavior over a longer term). This behavioral tendency is known as delay discounting and recent findings suggest that rates of delay discounting predict parents' use of harsh physical discipline. Existing research also indicates a strong link between steeper (more problematic) rates of delay discounting and the severity of alcohol and illicit drug use across the lifespan. Thus, delay discounting may represent a specific vulnerability underlying both harsh parenting and disordered substance use. The current project proposes to pilot and feasibility test an adapted episodic future thinking (EFT) intervention to target the reduction of parenting-related delay discounting and examine its effects on parenting practices among families in a residential substance use treatment setting. The intervention will be delivered by peer recovery coaches who are already employed in the center.

ELIGIBILITY:
Inclusion Criteria:

* Parent of child between 6-10 years of age
* Able to provide informed consent and take part in all study procedures in English
* Have current diagnosis of SUD
* Currently reside with their child at least 50% of the time
* Be willing to receive daily postcards

Exclusion Criteria:

* Active suicidality/homicidally
* Active bipolar disorder, schizophrenia, or psychosis.
* Only one parent-child dyad from each family.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Felton, PhD, Principal Investigator — Henry Ford Health
Locations (1):
- Odyssey Village, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staton-Tindall M, Sprang G, Clark J, Walker-Barnes R, Craig CD. Caregiver Substance Use and Child Outcomes: A Systematic Review. Journal of Social Work Practice in the Addictions. 2013;13(1):6-31. doi:10.1080/1533256X.2013.752272
- [Background] Committee on Child Maltreatment Research, Policy, and Practice for the Next Decade: Phase II; Board on Children, Youth, and Families; Committee on Law and Justice; Institute of Medicine; National Research Council; Petersen AC, Joseph J, Feit M, editors. New Directions in Child Abuse and Neglect Research. Washington (DC): National Academies Press (US); 2014 Mar 25. Available from http://www.ncbi.nlm.nih.gov/books/NBK195985/ PMID 24757747
- [Background] Herrenkohl RC, Herrenkohl EC, Egolf BP. Circumstances surrounding the occurrence of child maltreatment. J Consult Clin Psychol. 1983 Jun;51(3):424-31. doi: 10.1037//0022-006x.51.3.424. No abstract available. PMID 6863704
- [Background] Whipple EE, Richey CA. Crossing the line from physical discipline to child abuse: how much is too much? Child Abuse Negl. 1997 May;21(5):431-44. doi: 10.1016/s0145-2134(97)00004-5. PMID 9158904
- [Background] Alati R, Baker P, Betts KS, Connor JP, Little K, Sanson A, Olsson CA. The role of parental alcohol use, parental discipline and antisocial behaviour on adolescent drinking trajectories. Drug Alcohol Depend. 2014 Jan 1;134:178-84. doi: 10.1016/j.drugalcdep.2013.09.030. PMID 24479151
- [Background] Young NK, Boles SM, Otero C. Parental substance use disorders and child maltreatment: overlap, gaps, and opportunities. Child Maltreat. 2007 May;12(2):137-49. doi: 10.1177/1077559507300322. PMID 17446567
- [Background] Reynolds B. A review of delay-discounting research with humans: relations to drug use and gambling. Behav Pharmacol. 2006 Dec;17(8):651-67. doi: 10.1097/FBP.0b013e3280115f99. PMID 17110792
- [Background] Bickel WK, Marsch LA. Toward a behavioral economic understanding of drug dependence: delay discounting processes. Addiction. 2001 Jan;96(1):73-86. doi: 10.1046/j.1360-0443.2001.961736.x. PMID 11177521
- [Background] Amlung M, Vedelago L, Acker J, Balodis I, MacKillop J. Steep delay discounting and addictive behavior: a meta-analysis of continuous associations. Addiction. 2017 Jan;112(1):51-62. doi: 10.1111/add.13535. Epub 2016 Sep 1. PMID 27450931
- [Background] MacKillop J, Amlung MT, Few LR, Ray LA, Sweet LH, Munafo MR. Delayed reward discounting and addictive behavior: a meta-analysis. Psychopharmacology (Berl). 2011 Aug;216(3):305-21. doi: 10.1007/s00213-011-2229-0. Epub 2011 Mar 4. PMID 21373791
- [Background] Felton JW, Collado A, Ingram K, Lejuez CW, Yi R. Changes in delay discounting, substance use, and weight status across adolescence. Health Psychol. 2020 May;39(5):413-420. doi: 10.1037/hea0000833. Epub 2020 Jan 9. PMID 31916829
- [Background] Milligan K, Meixner T, Tremblay M, Tarasoff LA, Usher A, Smith A, Niccols A, Urbanoski KA. Parenting Interventions for Mothers With Problematic Substance Use: A Systematic Review of Research and Community Practice. Child Maltreat. 2020 Aug;25(3):247-262. doi: 10.1177/1077559519873047. Epub 2019 Oct 14. PMID 31610688
- [Background] Neger EN, Prinz RJ. Interventions to address parenting and parental substance abuse: conceptual and methodological considerations. Clin Psychol Rev. 2015 Jul;39:71-82. doi: 10.1016/j.cpr.2015.04.004. Epub 2015 Apr 24. PMID 25939033
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] Liu L, Feng T, Chen J, Li H. The value of emotion: how does episodic prospection modulate delay discounting? PLoS One. 2013 Nov 28;8(11):e81717. doi: 10.1371/journal.pone.0081717. eCollection 2013. PMID 24312341
- [Background] Peters J, Buchel C. Episodic future thinking reduces reward delay discounting through an enhancement of prefrontal-mediotemporal interactions. Neuron. 2010 Apr 15;66(1):138-48. doi: 10.1016/j.neuron.2010.03.026. PMID 20399735
- [Background] Lin H, Epstein LH. Living in the moment: effects of time perspective and emotional valence of episodic thinking on delay discounting. Behav Neurosci. 2014 Feb;128(1):12-9. doi: 10.1037/a0035705. PMID 24512061

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Episodic Future Thinking
Started | 38 (20 adults, 18 children)
Completed Baseline Questionnaire | 18
Completed Parent Intervention | 15
Completed Parent-Child Interaction (PCI) | 13
Completed | 30
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Population: Analyses of self-reported outcomes include only (n=15) parents who completed baseline and post-intervention. Additionally, only a subset of parents received the 5-trial adjusting measure. Only parent-child dyads that completed both the baseline and post-intervention parent-child interactions (n=6) were included in DPICS analyses.
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic data reported separately for parent and child participants.
  years
    Adult Participants: number analyzed (Participants) | 20
    Adult Participants | 37.6 (5.7)
    Child Participants: number analyzed (Participants) | 18
    Child Participants | 7.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographic data presented separately for parent and child participants.
  Participants
    Parent participants: number analyzed (Participants) | 20
    Parent participants: Female | 11
    Parent participants: Male | 9
    Child participants: number analyzed (Participants) | 18
    Child participants: Female | 14
    Child participants: Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic data reported separately for parent and child participants.
  Participants
    Parent participants: number analyzed (Participants) | 20
    Parent participants: Hispanic or Latino | 3
    Parent participants: Not Hispanic or Latino | 17
    Parent participants: Unknown or Not Reported | 0
    Child participants: number analyzed (Participants) | 18
    Child participants: Hispanic or Latino | 1
    Child participants: Not Hispanic or Latino | 17
    Child participants: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic data reported separately for parent and child participants.
  Participants
    Parent Participants: number analyzed (Participants) | 20
    Parent Participants: American Indian or Alaska Native | 00
    Parent Participants: Asian | 0
    Parent Participants: Native Hawaiian or Other Pacific Islander | 1
    Parent Participants: Black or African American | 4
    Parent Participants: White | 14
    Parent Participants: More than one race | 0
    Parent Participants: Unknown or Not Reported | 1
    Child Participants: number analyzed (Participants) | 18
    Child Participants: American Indian or Alaska Native | 0
    Child Participants: Asian | 0
    Child Participants: Native Hawaiian or Other Pacific Islander | 1
    Child Participants: Black or African American | 5
    Child Participants: White | 11
    Child Participants: More than one race | 1
    Child Participants: Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Delay Discounting 5 Trial Adjusted Measure
Description: The 5-Trial Adjusting Delay (Temporal Discounting) Task is a computer based system which uses an adjusting algorithm to determine the amount of immediately available money that is equivalent to a large sum that is delayed by seven discrete durations of time presented in a randomized order (i.e., 1 day, 1 week, 1 month, 6 months, 1 year, 5 years, and 25 years). The length of delay is titrated based on participants' responses to previous items to determine an "indifference point" (the point at which the sums of money are perceived as equal). This is then converted to a k-value and logarithmically transformed to ensure the values are normally distributed, making them unbounded by min and max values. Higher k-values indicate a greater preference for immediate rewards. Change in Delay Discounting is evaluated by comparing baseline k-value scores with scores at the intervention (approximately 1 week after baseline) and the post-intervention assessment (approximately 4 weeks after baseline).
Time Frame: Baseline and 4 weeks
Population: Participants included in analyses were those who completed the measure at both baseline and 4 weeks post.
Measure: Mean (Standard Deviation); unit: log (k)
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 11
log (k)
  Delay discounting (k-value) at baseline | -3.87 (3.81)
  Delay discounting (k-value) at follow-up | -5.03 (2.38)
Statistical Analysis 1: Comparison: Episodic Future Thinking; A single-sided paired-samples t-test comparing k-values at baseline to k-values at follow-up (approximately 4 weeks after baseline assessment) was examined. Given that k-values are typically skewed (and to be consistent with the existing literature) we used a log-k as our outcome variable; Test type: Superiority; p = .124, t-test, 1 sided; No adjustments were made. DF = 10; Mean Difference (Final Values) = 1.24

2. Primary Outcome: Change in Consideration of Future Consequences Scale - Parenting Adapted
Description: The Consideration of Future Consequences Scale-Parenting Adapted (CFCS-14-PA) is a 14-item self-report questionnaire composed of two subscales reflecting either immediate or future orientation related to parents interactions with their children. Items range from "not at all like me" (1) to "very much like me" (5) and are summed to create a total score with higher values reflecting greater future orientation. Scores range from 14 to 70. Change in CFCS-14-PA score is measured by comparing scores at the post-intervention assessment (approximately 4 weeks after baseline) with baseline scores.
Time Frame: Baseline, 4 weeks
Population: All parent participants who completed baseline and follow-up assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 15
score on a scale
  CFCS-14-PA Total Score at Baseline | 54.93 (6.08)
  CFCS-14-PA Total Score at Follow-Up | 53.80 (7.82)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Changes in consideration of future consequences (parenting) was evaluated using one-sided paired samples t-tests; Test type: Superiority; p = .219, t-test, 1 sided; No adjustments were made. DF = 14; Mean Difference (Final Values) = 1.13

3. Secondary Outcome: Change in Dyadic Parent-Child Interaction Coding System Scores
Description: Parents and their children will complete a 20-minute interaction task, including 5 min. of free play, a 10 min. "homework" task, and a 5 min. clean up task. Interactions are recorded and coded using the Dyadic Parent-Child Interaction Coding System (DPICS), measuring the quality of parent and child interactions. The task is coded for 7 subscales, yielding 2 composite scores: positive parenting (a sum of: unlabeled praise, labeled praise, positive touch, reflection, and behavior description) and negative parenting (a sum of: negative talk and negative touch). Each instance of a behaviors described in the subscale (e.g., a parent giving unlabeled praise) is coded as one "point," which are summed into a subscale (no max or min values). Higher values indicate greater positive or negative parenting. Change in positive parenting and negative parenting scores will be calculated by comparing baseline scores with scores at the post-intervention sessions (approximately 4 weeks after baseline).
Time Frame: Baseline, 4 weeks
Population: Analyses included 6 parent-child dyads who completed both the pre- and post-intervention parent-child interaction task.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 6
score on a scale
  Positive Parenting Composite at Baseline | 4.83 (2.48)
  Negative Parenting at Baseline | 3.17 (4.07)
  Positive Parenting Composite at Follow-Up | 4.83 (3.60)
  Negative Parenting at Follow-Up | 5.17 (1.94)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Performed a one-sided paired samples t-test examining changes in both positive parenting; Test type: Superiority; p = .50, t-test, 1 sided; No adjustments were made. DF = 5; Mean Difference (Final Values) = 0.00
Statistical Analysis 2: Comparison: Episodic Future Thinking; Used a one-sided paired samples t-test to examine changes in negative parenting; Test type: Superiority; p = .187, t-test, 1 sided; Mean Difference (Final Values) = -1.0

4. Secondary Outcome: Change in Alabama Parenting Questionnaire Scores
Description: The Alabama Parenting Questionnaire (APQ) is a 42-item self-report measure of parenting behaviors which yields five subscales: (1) positive involvement with children (range 10-50, higher = more involvement), (2) use of positive parenting strategies (range 6-30, higher = more positive strategies), (3) poor parental monitoring/supervision (range 10-50, higher = worse supervision), (4) inconsistent discipline (range 6-30, higher = more inconsistent discipline), and (5) use of corporal punishment (range 3-15, higher = more corporal punishment). Items are summed to create subscale scores. Change in each of the five APQ subscale scores will be measured by comparing post-intervention scores (approximately 4 weeks after baseline) with baseline scores.
Time Frame: Baseline, 4 weeks
Population: All parents who completed the APQ at baseline and post-intervention were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Episodic Future Thinking
Number analyzed (Participants) | 13
score on a scale
  Involved Parenting at Baseline | 38.93 (6.08)
  Positive Parenting at Baseline | 26.5 (2.79)
  Poor Parental Monitoring at Baseline | 15.22 (4.54)
  Inconsistent Parenting at Baseline | 15.14 (3.84)
  Corporal Punishment at Baseline | 5.21 (1.93)
  Involved Parenting at Follow-Up | 38.94 (6.88)
  Positive Parenting at Follow-Up | 25.71 (3.38)
  Poor Parental Monitoring at Follow-Up | 16.43 (4.80)
  Inconsistent Parenting at Follow-Up | 15.66 (3.96)
  Corporal Punishment at Follow-Up | 5.07 (1.54)
Statistical Analysis 1: Comparison: Episodic Future Thinking; Examined changes in parental involvement using a paired-samples t-test; Test type: Superiority; p = .498, t-test, 1 sided; Mean Difference (Final Values) = -.01
Statistical Analysis 2: Comparison: Episodic Future Thinking; Examined changes in positive parenting using paired samples t-tests; Test type: Superiority; p = .108, t-test, 1 sided; Mean Difference (Final Values) = 1.301
Statistical Analysis 3: Comparison: Episodic Future Thinking; Examined changes in parental monitoring using a paired samples t-test; Test type: Superiority; p = .145, t-test, 1 sided; Mean Difference (Final Values) = -1.01
Statistical Analysis 4: Comparison: Episodic Future Thinking; Examined changes in inconsistent parenting using a paired samples one-sided t-test; Test type: Superiority; p = .252, t-test, 1 sided; Mean Difference (Final Values) = -.688
Statistical Analysis 5: Comparison: Episodic Future Thinking; Examined changes in corporal punishment using a paired samples one-tailed t-test; Test type: Superiority; p = .382, t-test, 1 sided; Mean Difference (Final Values) = .306

ADVERSE EVENTS:
Time Frame: Participants were involved in the study for approximately four weeks from consent to follow-up period.
Arm/Group | Episodic Future Thinking
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05229120/Prot_SAP_000.pdf